CLINICAL TRIAL: NCT02634957
Title: Impact of Duration Of Absolute Voice Rest on Voice Outcome After Phonomicrosurgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to change in available resources
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Libby Smith DO, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO15120009
Record Dates: First submitted 2015-12-11; First posted 2015-12-18 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Benign Neoplasm of True Vocal Cords
Keywords: phonomicrosurgery; benign vocal fold lesions; voice rest; vhi-10; CPP

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 day absolute voice rest (Experimental): participants would begin initiation of voice/speaking 3 days post phonomicrosurgery for benign vocal fold lesions
  Interventions: Behavioral: absolute voice rest
- 7 day absolute voice rest (Experimental): participants would begin initiation of voice/speaking 7 days post phonomicrosurgery for benign vocal fold lesions
  Interventions: Behavioral: absolute voice rest

INTERVENTIONS:
Behavioral: absolute voice rest — absolute voice rest is the complete elimination of any vocalization (no sounds, speaking or whispering)

SUMMARY:
Absolute voice rest is commonly prescribed after vocal fold surgery, also known as phonomicrosurgery, for benign vocal fold lesions. This is thought to decrease scarring of vocal folds, which could result in increasing tissue stiffness and limitations in optimal vocal outcome. Unfortunately there is no standardized protocol as to how long patients should rest their voice after phonomicrosurgery. To date, there are no studies in the literature directly comparing the impact of short-term and long-term voice rest on vocal fold healing and voice outcome after phonomicrosurgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether 3 days versus 7 days of absolute voice rest will result in different voice outcomes in patients who have undergone phonomicrosurgery for benign vocal fold lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with benign mid membranous vocal fold lesions such as the following:

   1. Polyps
   2. Cysts
   3. Sub-epithelial fibrous mass
2. Undergoing elective phonomicrosurgery for vocal fold lesions, which involves microflap excision +/- truncation +/- steroid injection into the vocal folds.
3. Age 18 and older

Exclusion Criteria:

Patients with any of the following will be excluded from the study:

1. Reinke's edema
2. Active smokers
3. Ligamentous mid membranous vocal fold lesions
4. RRP (Recurrent Respiratory Papillomatosis)
5. Dysplasia
6. CIS (Carcinoma-in-situ)
7. SCC (squamous cell carcinoma)
8. Extent of surgery exceeds what is mentioned in the inclusion criteria (e.g., CO2 laser, balloon dilatation, vocal fold augmentation in addition to phonomicrosurgery)
9. Previous vocal fold surgery
10. Systemic steroids
11. History of systemic illness that could affect wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index - 10 | 3 months post op
Voice Handicap Index - 10 | 1 month post op

SECONDARY OUTCOMES:
Cepstral Peak Prominence (CPP) | 1 month and 3 months post op
Average phonatory airflow in all voiced sentence | 1 month and 3 months post op
video stroboscopy findings | 1 month and 3 months post op

CONTACTS AND LOCATIONS:
Overall Officials: Libby Smith, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified information with outside collaborators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: information may be shared during and after collection for the purpose of analysis
Access Criteria: if not part of original IRB, sharing will only occur if there is a data use agreement executed.